CLINICAL TRIAL: NCT04055532
Title: Biomarkers in Neurodegenerative Diseases
Status: Withdrawn | Type: Observational
Why Stopped: Lack of regulatory approval
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00007108
Record Dates: First submitted 2019-08-12; First posted 2019-08-13 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Mild Cognitive Impairment (MCI); Alzheimer Disease (AD); Dementia With Lewy Bodies (DLB); Frontotemporal Lobar Degeneration (FTLD); Parkinsons Disease With Dementia (PDD); Transient Epileptic Amnesia (TEA); Temporal Lobe Epilepsy (TLE); Spinocerebellar Ataxias (SCA); HIV Associated Neurocognitive Disorder (HAND); Amyotrophic Lateral Sclerosis (ALS); Primary Lateral Sclerosis (PLS)
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Lewy Body Disease; Frontotemporal Lobar Degeneration; Epilepsy, Temporal Lobe; Spinocerebellar Ataxias; Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- Mild Cognitive Impairment
  Interventions: Other: Neuraceq
- Alzheimer's Disease
  Interventions: Other: Neuraceq
- Dementia with Lewy Bodies
  Interventions: Other: Neuraceq
- Frontotemporal Lobar Dementia
  Interventions: Other: Neuraceq
- Parkinson's Disease with Dementia
  Interventions: Other: Neuraceq
- Transient Epileptic Amnesia
  Interventions: Other: Neuraceq
- Temporal Lobe Epilepsy
  Interventions: Other: Neuraceq
- Spinocerebellar Ataxia
  Interventions: Other: Neuraceq
- HIV-Associated Neurocognitive Disorder
  Interventions: Other: Neuraceq
- Amyotrophic Lateral Sclerosis
  Interventions: Other: Neuraceq
- Primary Lateral Sclerosis
  Interventions: Other: Neuraceq

INTERVENTIONS:
Other: Neuraceq — Neuraceq is a radioactive isotope used for Amyloid-beta-PET/CT scans.

SUMMARY:
The general purpose of this observational study is to examine biomarkers associated with the pathology of neurodegenerative diseases to potentially develop novel therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MCI, AD, DLB, FTLD, PDD, TEA, TLE, SCA, HAND, ALS, PLS, or normal control.
2. Age 18 or older
3. Reliable informant with frequent contact with participant
4. Mini Mental State Exam (MMSE) ≥15 AND/OR Clinical Dementia Rating (CDR) less than 2
5. Able to undergo extensive psychometric testing

Exclusion Criteria:

1. Any conditions that could account for cognitive deficits in addition to a neurodegenerative disease, including but not limited to:

   * Past or present diagnosis of Korsakoff's syndrome
   * Alcohol or substance abuse preceding dementia & still present within 5 years of onset
   * Present untreated vitamin B12 or folate deficiency
   * Present untreated hypothyroidism
   * Past or present head trauma with persistent deficits
   * Present untreated syphilis
   * Past or present multiple sclerosis or another neuro-inflammatory disorder
   * Past or present vascular or multi-infarct dementia
   * Past or present diagnosis of huntington's disease
   * Past or present normal pressure hydrocephalus
   * Past or present central nervous system (CNS) lesions deemed to be clinically significant
   * Unresolved or present subdural hematoma
   * Past or present Ischemic Vascular Dementia
   * Past or present intracerebral hemorrhage
   * Present systematic liver disease
   * Present renal insufficiency requiring dialysis
   * Present encephalitis or meningitis
   * Present anxiety disorder (not due to dementia and requiring medication more than 3x per week)
   * Present severe periventricular white matter disease or greater than grade 4 white matter lesions
   * Present lacunar infarcts deemed to clinically significant
   * Present cortical stroke
   * Present respiratory condition requiring oxygen
2. Present significant systemic medical illness, such as cancer requiring chemotherapy or end stage cardiac insufficiency
3. Present inability to safely scan in an MRI
4. Present pregnancy or lactation - Female participants will be asked to confirm that they are not pregnant and do not plan to become pregnant.
5. Present current medication likely to affect CNS functions:

   * Benzodiazepines (no triazolam, but other short-acting benzodiazepines are OK)
   * Antidepressant therapy with amitriptyline or doxepin or tx not stable during past year
   * Neuroleptics in the phenothiazine and haloperidol families (atypicals OK)
   * Narcotics (codeine is OK, but hold 24 hours before neuropsychological testing)
   * Anti-seizure medication outside of therapeutic ranges
   * Antihistamines (> 3x per week; hold 24 hours before neuropsychological testing)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Adults lacking capacity to consent and/or adults with diminished capacity to consent, including, but not limited to, those with acute medical conditions, psychiatric disorders, neurologic disorders, developmental disorders, and behavioral disorders.
  * Individual or group with a serious health condition for which there are no satisfactory standard treatments.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Performance on Batteries of Cognitive Tests | 2-5 Years
  Performance on batteries of cognitive tests as measured by the Modified Autobiographical Memory Interview (MAMI), Stroop Test, CDR-SOB, Spontaneous Speech Test, and the Neuropsychological Battery from the Uniform Data Set.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Vossel, MD, MSc, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided